CLINICAL TRIAL: NCT06190821
Title: Hydrodissection of the Hepatoduodenal Ligament
Acronym: Duodenal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8695
Record Dates: First submitted 2022-09-06; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Lesions
Keywords: hepatic lesions; liver lesions; duodenum; hepato duodenal ligament

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous treatment of liver lesions adjacent to the duodenum exposes the duodenum to the risk of thermal injury, limiting removal and oncologic outcome. In this study the investigators investigate the feasibility of hepato duodenal ligament dissection in the percutaneous treatment of liver lesions adjacent to the duodenum.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years of age)
* Subject who underwent percutaneous ablation of primary or secondary liver lesions at HUS that required per-procedure hepatoduodenal ligament hydrodissection in the interventional imaging department of the New Civil Hospital from January 2019 to July 2022.
* Subject who has not expressed opposition to the reuse of their data for the purpose of this research.

Exclusion Criteria:

- Opposition to the reuse of his/her data for the purpose of scientific research.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years of age) who underwent percutaneous ablation of primary or secondary liver lesions at HUS that required per-procedure hepatoduodenal ligament hydrodissection in the interventional imaging department of the New Civil Hospital from January 2019 to July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the hepatoduodenal ligament dissection in the percutaneous treatment of liver lesions adjacent to the duodenum | Files analysed retrospectively from January 01, 2019 to July 31, 2022 will be examined
  This study is retrospective

CONTACTS AND LOCATIONS:
Locations (1):
- Service Imagerie interventionnelle oncologique et viscérale - CHU de Strasbourg - France, Strasbourg, France